CLINICAL TRIAL: NCT03441061
Title: Phase II Study of Inotuzumab Ozogamicin in Patients With B-Cell Lineage Acute Lymphocytic Leukemia With Positive Minimal Residual Disease
Brief Title: Inotuzumab Ozogamicin in Treating Patients With B-cell Acute Lymphocytic Leukemia With Positive Minimal Residual Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0921; NCI-2018-00936 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0921 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia; Recurrent B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (inotuzumab ozogamicin) (Experimental): Patients receive inotuzumab ozogamicin IV over 1 hour on days 1 and 8. Treatment repeats every 21-28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Inotuzumab Ozogamicin

INTERVENTIONS:
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294

SUMMARY:
This phase II trial studies how well inotuzumab ozogamicin works in treating patients with B-cell acute lymphocytic leukemia with positive minimal residual disease. Inotuzumab ozogamicin is a monoclonal antibody called inotuzumab linked to a toxic agent called ozogamicin. Inotuzumab ozogamicin attaches to B cell-specific CD22 cancer cells in a targeted way and kills them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the clinical efficacy of inotuzumab ozogamicin in patients B-cell acute lymphoblastic leukemia (ALL) in complete morphologic remission with positive minimal residual disease (MRD) in terms of relapse-free survival (RFS).

SECONDARY OBJECTIVE:

I. To evaluate other efficacy endpoints such as overall survival and MRD negativity rate by flow cytometry and/or polymerase chain reaction (PCR) overall and after the first cycle, as well as safety of inotuzumab ozogamicin in this setting.

OUTLINE:

Patients receive inotuzumab ozogamicin intravenously (IV) over 1 hour on days 1 and 8. Treatment repeats every 21-28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 day and then periodically every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-lineage ALL in hematologic complete remission (CR) with molecular failure (ie, had never achieved an MRD-negativity status before inotuzumab ozogamicin) or had a molecular relapse (ie, became MRD positive after having been MRD negative) starting at any time point after 3 months of frontline therapy. Molecular disease or minimal residual disease is defined by any level of measurable residual disease identified by multicolor flow cytometry, PCR and/or next-generation sequencing (NGS).
* Patients with B-lineage ALL in at least marrow CR in salvage 1 and beyond with MRD failure at any time point after 1 month of salvage therapy are allowed, including patients who received prior allogeneic stem cell transplantation.
* Patients with Ph+ ALL can be enrolled in CR1 or CR2 and beyond. A TKI will be added at the discretion of the treating physician. MRD for these patients will be defined by either 1.) a ratio of BCR-ABL1 to ABL1 by PCR of ≥ 0.01% according to the International Scale for patients with p210 transcript or a ratio of BCR-ABL1 to ABL1 by PCR of ≥ 0.01% for patients with non-p210 transcripts, or 2.) detectable MRD at any level of measurable residual disease identified by multicolor flow cytometry and/or by NGS.
* Performance status of 0, 1, or 2
* Creatinine clearance >= 15 ml/min
* Bilirubin < 1.5 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 X ULN
* No active or co-existing malignancy with life expectancy less than 12 months

Exclusion Criteria:

* Pregnant or nursing women
* Known to be human immunodeficiency virus positive (HIV+)
* Active and uncontrolled disease/infection as judged by the treating physician
* Unable or unwilling to sign the consent form
* Active central nervous system (CNS) or extramedullary disease
* Monoclonal antibodies therapy within 2 weeks before study entry
* Radiotherapy or cancer chemotherapy (except for intrathecal prophylaxis and/or low-dose maintenance therapy such as vinca alkaloids, mercaptopurine, methotrexate, steroids) or any investigational drug within 2 weeks before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | Up to 4 years

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 4 years
  Will continuously monitor treatment-related toxicities using the Bayesian approach of Thall, Simon, Estey. For the purpose of toxicity monitoring, toxicities are defined as any treatment-related grade 3 or 4 non-hematologic adverse events occurring any time during the trial.
Overall survival | Up to 4 years
Minimal residual disease (MRD) negativity rate | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Zhao Y, Short NJ, Kantarjian HM, Chang TC, Ghate PS, Qu C, Macaron W, Jain N, Thakral B, Phillips AH, Khoury J, Garcia-Manero G, Zhang W, Fan Y, Yang H, Garris RS, Nasr LF, Kriwacki RW, Roberts KG, Konopleva M, Jabbour EJ, Mullighan CG. Genomic determinants of response and resistance to inotuzumab ozogamicin in B-cell ALL. Blood. 2024 Jul 4;144(1):61-73. doi: 10.1182/blood.2024023930. PMID 38551807
- [Derived] Jabbour E, Haddad FG, Short NJ, Senapati J, Jain N, Sasaki K, Jorgensen J, Wang SA, Alvarado Y, Wang X, DiNardo C, Masarova L, Kadia T, Garris RS, Ravandi F, Kantarjian H. Phase 2 study of inotuzumab ozogamicin for measurable residual disease in acute lymphoblastic leukemia in remission. Blood. 2024 Feb 1;143(5):417-421. doi: 10.1182/blood.2023022330. PMID 37879077
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- See also: MD Anderson Cancer Center — https://www.mdanderson.org/